CLINICAL TRIAL: NCT06891859
Title: Investigation of the Relationship Between Static and Dynamic Balance Performance and Temporomandibular Dysfunction Symptoms in Healthy Adults
Brief Title: Temporomandibular Disorders and Balance Performance
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Mert Durukan, Graduate Assistant, Bandırma Onyedi Eylül University
Other Study IDs: 2024 -31
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-08

CONDITIONS: University Students
Keywords: head posture; masseter; body balance; temporomandibular joint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to investigate the relationship of the temporomandibular joint with head posture, pressure pain threshold, and body balance.

DETAILED DESCRIPTION:
This cross-sectional study was conducted on university students aged 18-30 between April 2024 and December 2024. In the evaluation of the students, the Fonseca Anamnestic Questionnaire was used for temporomandibular joint dysfunction, the Research Diagnostic Criteria for Temporomandibular Disorders Examination Form was used for maximum pain-free mouth opening, presence of sound in temporomandibular joint movements, and palpation parameters of the temporomandibular joint and surrounding muscles. An algometer device was used for pressure pain threshold measurement, a goniometer for head-neck posture, EMG for measuring the activation of the masseter muscle, and the Korebalance Premier-19 device for static and dynamic body balance measurement.

ELIGIBILITY:
Inclusion Criteria:

* Must be a student at Bandırma Onyedi Eylül University
* Must be willing to participate in the study
* Aged between 18-30

Exclusion Criteria:

* Individuals who have undergone masseter botox treatment
* Individuals diagnosed with temporomandibular joint disorders and/or bruxism
* Individuals with musculoskeletal problems showing evidence of specific pathological conditions, such as fractures or rheumatoid diseases related to the lower extremities, spine, and/or temporomandibular joint
* Individuals who have undergone any surgery related to the lower extremities, spine, and/or temporomandibular joint
* Individuals who have received physical therapy related to the lower extremities, spine, and/or temporomandibular joint within the last six months
* Individuals diagnosed with psychiatric disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University students
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Data Form | February 2024 and June 2024
  Through this form, fundamental information such as the participants' age, height, body weight, sex, educational status, occupation, and marital status was recorded, along with their medical history, current medication use, past surgical interventions, and whether any treatment or intervention related to the temporomandibular joint (TMJ) had been performed within the last six months.
Pressure pain threshold | February 2024 and June 2024
  Pressure pain threshold The pressure pain threshold measurement was conducted on the masseter muscles using an algometer.
Numerical Pain Scale (NPS) Assessment | February 2024 and June 2024
  This scale ranges from 0 to 10, where patients indicate their pain level by selecting a number within the range of "0 - no pain" to "10 - worst possible pain" to describe the intensity of their experienced pain.
Forward head posture | February 2024 and June 2024
  It was evaluated using the craniovertebral angle (CVA) method. The craniovertebral angle is defined as the angle formed between the horizontal line and the line connecting the tragus of the ear to the spinous process of the seventh cervical vertebra.
Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) | February 2024 and June 2024
  This form consists of criteria used for the diagnosis of commonly encountered temporomandibular disorders (TMD). Based on the results of the form, participants can be diagnosed with one or more conditions such as myofascial pain, osteoarthritis, arthralgia, disc displacement, and arthritis.
  DC/TMD consists of two main sections. The first section includes criteria for diagnosing disorders related to the masticatory muscles and the temporomandibular joint (TMJ). The second section allows for a comprehensive assessment of pain and the individual's psychosocial status by evaluating factors such as pain intensity, pain-related disabilities, depression, and somatization.
Maximum pain-free mouth opening | February 2024 and June 2024
  The maximum pain-free mouth opening was recorded using a 10 cm ruler.
Fonseca's Anamnestic Questionnaire | February 2024- June 2024
  Fonseca's Anamnestic Questionnaire (FAQ) was used for TMJ dysfunction. The FAQ has a multi-factor evaluation structure. The questionnaire consists of ten questions about pain in TMJ, head, and joints, with answer options of "No, Sometimes and Yes." A score of 25 and above was accepted as the presence of TMD.
Muscle Activation Assessment | February 2024 and June 2024
  In our study, a four-channel Neurotrac MyoPlus Pro 4 surface EMG biofeedback device was used to assess muscle activation. Participants sat in an upright position with standardized posture, and EMG signals were recorded from the bilateral masseter muscles using self-adhesive electrodes. EMG signals were recorded using self-adhesive electrodes measuring 2.5 cm × 2.5 cm. The electrodes were placed bilaterally on the masseter muscles, with an inter-electrode distance of 10 mm. Before normalization, maximum voluntary isometric contraction (MVIC) levels were recorded. Participants performed three five-second maximal clenching trials with one-minute rest intervals. After the MVIC measurement, bilateral masseter muscle activation was recorded again via EMG during balance assessments. Muscle activation during the task was analyzed using Neurotrac PC Software, and the results were reported as mean microvolt values and normalized data (%MVC).
Static and Dynamic Balance Assessment | February 2024 and June 2024
  The Korebalance Premier-19 device was used to measure postural imbalances through anterior-posterior and medial-lateral sway. Postural deviations were assessed using a total score, where higher scores indicated poorer balance.
  Static balance was tested with both eyes open and closed, with the device inflated to 6.0 PSI. Participants were instructed to maintain a stable posture and keep the "+" sign centered on the monitor. In the eyes-closed test, they adjusted their balance and position before the measurement began, followed by a five-second countdown, after which they attempted to maintain the same balance and position.
  Dynamic balance was assessed only with eyes open, with the device inflated to 5.0 PSI. Participants tracked a moving target without external support. Each balance assessment lasted 30 seconds per participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Bandirma Onyedi Eylul University, Balıkesir, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided